CLINICAL TRIAL: NCT06160089
Title: Effectiveness of Iso-inertial Resistance Training on the Muscle Power of the Lower Limbs, Physical Aptitude, and Risk of Falls in Physically Active Older Adults: a Randomised Controlled Trial
Brief Title: Effectiveness of Iso-inertial Resistance Training in Physically Active Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Aïda Cadellans-Arróniz, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FIS-2023-03
Record Dates: First submitted 2023-11-06; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Aged; Muscle Strength; Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a parallel group, randomized controlled trial (allocation ratio 1:1) with blinded outcome assessment where participants will be randomly assigned to one of the two study groups (iso-inertial or gravitational resistance training).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gravitational group (Active Comparator): Participants will have to perform a 6-week programme based on three exercises: front lunge, side lunge, and front lunge with hand grip pull, that will be the basis of each session. Exercices will be performed with the gravitational device.
  Interventions: Other: Gravitational training
- Isoinertial group (Experimental): Participants will have to perform a 6-week programme based on three exercises: front lunge, side lunge, and front lunge with hand grip pull, that will be the basis of each session. Exercices will be performed with the isoinertial device.
  Interventions: Other: Isoinertial training

INTERVENTIONS:
Other: Isoinertial training — For the front lunge and the front lunge with hand grip pull, the participant will be placed frontally on the training device (inertial). Whereas for the side lunge the participant will be placed sideways on the device (homolateral on the scrolling limb). For front and side lunge, a weight shift belt will be used, which will be placed on the waist. For the frontal lunge with hand grip pull, the grip is performed with the upper limb homolateral to the displaced lower limb. The volume and difficulty of execution of the exercises will increase over time. Investigators will instruct the participants to perform the exercises at a given intensity according to the Borg Rating of Perceived Exertion (RPE) scale. The intensity will increase throughout the training program.
  Arms: Isoinertial group
Other: Gravitational training — For the front lunge and the front lunge with hand grip pull, the participant will be placed frontally on the training device (gravitational). Whereas for the side lunge the participant will be placed sideways on the device (homolateral on the scrolling limb). For front and side lunge, a weight shift belt will be used, which will be placed on the waist. For the frontal lunge with hand grip pull, the grip is performed with the upper limb homolateral to the displaced lower limb. The volume and difficulty of execution of the exercises will increase over time. Investigators will instruct the participants to perform the exercises at a given intensity according to the Borg Rating of Perceived Exertion (RPE) scale. The intensity will increase throughout the training program.
  Arms: Gravitational group

SUMMARY:
Strength training is effective for promoting longevity. The iso-inertial training method is an innovative way to improve strength, but it is unclear whether it improves muscle power and functional variables that are key to develop activities of daily living. The purpose of this study is to conduct a randomised controlled trial at the gymnasium Espai Esport Wellness Center (Granollers) involving physically active older adults (age ≥60). Our goal is to evaluate the effectiveness of a 6-week iso-inertial strength program on the muscle power, physical fitness and risk of falls compared to executing that program with a traditional gravitational strength method. Providing older adults with new, effective methods to preserve their functional capacities is essential for longevity. Also, bringing them into an active environment could encourage a healthier lifestyle and reduce the risk of physical and mental diseases.

DETAILED DESCRIPTION:
With the progressive increase in life expectancy of the population, attention to ageing has gained special interest in recent years. Actions aimed at promoting healthy ageing in the older adults are key to slow down the physiological progressive loss in skeletal muscle mass, quality and function as the person ages. These losses affect the individual's ability to carry out activities of daily living. More concretely, the muscle strength and power are reduced during aging, which has a negative impact on the functional capacity and quality of life of older adults. In fact, recent research has identified a significant decrease in muscle strength of 1-1.5% each year from the age of 50. While the muscle strength is defined as the ability to generate intramuscular tension when facing a resistance, regardless of whether it generates movement, the muscle power is defined as the maximum amount of force one can generate during a specific movement at a specified velocity. Previous studies report that muscle power is diminished to a greater extent than strength over time. Muscle power is considered a predictor of functional capacity, as it is associated with activities of daily living such as climbing stairs, standing up from a chair or walking. This fact has justified the use of strength and power training in different studies that aim to prevent the risk of falls, improve the balance or the walking capacity in older adults.

Resistance training (RT) is one of the main strategies to prevent the decrease in functional capacities and has demonstrated its effectiveness in combating age-induced muscle atrophy (sarcopenia), risk of falls, and fragility. RT has also been shown to improve cardiovascular health. Regarding the types of RT, previous studies have noted statistically significant differences in favor of eccentric training, when comparing it with concentric RT. Specifically, it has been observed that eccentric training leads to higher peak strength with lower muscle activation and lower metabolic cost, increased muscle mass and higher jumping performance. Thus, the values of muscle strength and power resulting from an eccentric RT are physiologically superior to those obtained when performing concentric RT.

The most traditionally used RT method in the field of community health is the one known as gravitational, in which a resistance is opposed through free weights or by blocks or disks in cable machines. One of the main restrictions of this method is that the workload applied during the shortening-longing cycle of a repetition is limited to concentric muscle capacity and does not allow a progression of the eccentric workload. This fact limits the potential of this method for generating the improvements associated with eccentric training mentioned above. In contrast, the iso-inertial (ISI) training method is based on the application of resistance generated by an iso-inertial device, where the workload is provided by the inertia of a rotating mass. Unlike the gravitational system, the ISI method can provide a resistance workload in the eccentric phase that is proportional to the concentric phase. Thanks to that, high workloads can be applied for both phases. Another benefit of ISI method is that, when the load increases or the fatigue appears, only the execution speed is reduced but the execution is not interrupted .

Different studies show that eccentric overload training protocols (i.e., with a higher force in the eccentric phase of a repetition) improve muscle hypertrophy and power, as well as and neuromuscular functions. Because of its force-generating system, the ISI method is ideal for eccentric overload compared to gravitational systems, where eccentric overload can only be achieved with external assistance. Also, the ISI method allows a fluid movement compared to the interrupted movements of gravitational systems.

Recent studies have reported improvements in postural control or maximal isometric strength with ISI training in older adults. Also for metabolic variables such as lipid profile or maximum oxygen volume consumption . However, no study has been found that compares the effects of ISI and gravitational training on muscle power and other relevant functional variables in older adults. This is of critical importance because of the direct implications that the improvements of muscle power has on activities of the daily live.

The main objective of this study is to evaluate the effectiveness of an iso-inertial resistance training program on the eccentric muscle power of the lower limbs compared to the same program executed with gravitational resistance in physically active older adults. The secondary objectives are 1) to evaluate the effectiveness of an iso-inertial resistance training program on the concentric muscle power, physical fitness (balance, walking speed and functionality of the lower limbs), and risk of falls compared to the same program executed with gravitational resistance in physically active older adults, and 2) to assess the differences between men and women for the previous objectives.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 or more.
* Adults physically active. By "physically active" we consider that they are enrolled in the gymnasium Espai Esport Wellness Centre and that they make use of their facilities with varying frequency in the months prior to the start of the study.

Exclusion Criteria:

* Acute Osteoarticular injuries
* Acute musculoskeletal injuries
* Systemic diseases
* Neurodegenerative diseases

Ages: 57 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
Muscle power during the eccentric | Before the first training session and one week after the last training session
  Muscle power during the eccentric phase measured with both iso-inertial and gravitational devices, measured with a rotatory and a linear encoder (Chronojump Boscosystem®), respectively.

SECONDARY OUTCOMES:
Muscle power during the concentric | Before the first training session and one week after the last training session
  Muscle power during the concentric phase measured with both iso-inertial and gravitational devices (measured with the encoders mentioned above)
Balance | Before the first training session and one week after the last training session
  Tandem and semitandem test, measured in seconds
Risk of falls | Before the first training session and one week after the last training session
  Get up and go test, measured in seconds
Walking speed | Before the first training session and one week after the last training session
  4 meters walking test, measured in seconds
Lower limb functionality | Before the first training session and one week after the last training session
  5 times sit to stand test, measured in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided